CLINICAL TRIAL: NCT00023335
Title: TBTC Study 22: Efficacy and Safety of Once-Weekly Rifapentine and Isoniazid Compared to Efficacy and Safety of Once-Weekly Rifapentine and Isoniazid Compared to Twice-Weekly Rifampin and Isoniazid in the Continuation Phase of Therapy for Pulmonary Tuberculosis
Brief Title: TBTC Study 22: Efficacy of Once-Weekly Rifapentine and Isoniazid in Treatment of Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-1427; TBTC Study 22
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — rifapentine; Isoniazid

INTERVENTIONS:
Drug: Rifapentine
Drug: Isoniazid

SUMMARY:
Primary Objective: To compare, at the completion of the follow-up phase, the clinical and bacteriologic relapse rates associated with the two study regimens.

Secondary Objectives:

To compare the clinical and bacteriologic failure rates of the two study regimens at the completion of the study phase therapy.

To compare the clinical and bacteriologic response rates for the two study regimens among patients who began study phase therapy with signs and symptoms of tuberculosis or cultures positive for M. tuberculosis.

To compare the toxicity associated with the two study regimens by comparing discontinuation rates due to adverse events and occurrence rates of signs and symptoms associated with adverse events during study phase therapy.

To compare mortality rates of the two study regimens. To compare the rates of completion of therapy within 22 weeks for the two study regimens.

To compare the rate of development of drug-resistant tuberculosis in the two study regimens among study patients classified as treatment failures or relapses.

To compare all of the above performance characteristics for the two study regimens in a small subset of HIV seropositive patients.

To compare attitudes and beliefs about participation in this study between patients who complete study therapy and those who fail to complete study therapy.

ELIGIBILITY:
* Culture-positive, drug-susceptible pulmonary tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 1995-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Background] Weiner M, Burman W, Vernon A, Benator D, Peloquin CA, Khan A, Weis S, King B, Shah N, Hodge T; Tuberculosis Trials Consortium. Low isoniazid concentrations and outcome of tuberculosis treatment with once-weekly isoniazid and rifapentine. Am J Respir Crit Care Med. 2003 May 15;167(10):1341-7. doi: 10.1164/rccm.200208-951OC. Epub 2003 Jan 16. PMID 12531776
- [Background] Benator D, Bhattacharya M, Bozeman L, Burman W, Cantazaro A, Chaisson R, Gordin F, Horsburgh CR, Horton J, Khan A, Lahart C, Metchock B, Pachucki C, Stanton L, Vernon A, Villarino ME, Wang YC, Weiner M, Weis S; Tuberculosis Trials Consortium. Rifapentine and isoniazid once a week versus rifampicin and isoniazid twice a week for treatment of drug-susceptible pulmonary tuberculosis in HIV-negative patients: a randomised clinical trial. Lancet. 2002 Aug 17;360(9332):528-34. doi: 10.1016/s0140-6736(02)09742-8. PMID 12241657
- [Background] Vernon A, Burman W, Benator D, Khan A, Bozeman L. Acquired rifamycin monoresistance in patients with HIV-related tuberculosis treated with once-weekly rifapentine and isoniazid. Tuberculosis Trials Consortium. Lancet. 1999 May 29;353(9167):1843-7. doi: 10.1016/s0140-6736(98)11467-8. PMID 10359410
- [Derived] Yamshchikov AV, Kurbatova EV, Kumari M, Blumberg HM, Ziegler TR, Ray SM, Tangpricha V. Vitamin D status and antimicrobial peptide cathelicidin (LL-37) concentrations in patients with active pulmonary tuberculosis. Am J Clin Nutr. 2010 Sep;92(3):603-11. doi: 10.3945/ajcn.2010.29411. Epub 2010 Jul 7. PMID 20610636
- See also: Click here for more information about the Tuberculosis Trials Consortium (TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/